CLINICAL TRIAL: NCT06537232
Title: A Randomized Crossover-Controlled Trial Investigating the Epigenetic Impact of a Greens-Based Supplement in Adults
Brief Title: Greens-Based Crossover Trial to Improve Epigenetic Aging in Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Collaborators: Brickhouse Nutrition (Unknown)
Responsible Party: Principal Investigator, Andrew Fruge, Associate Professor, Auburn University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AUBHG 24
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Aging
Keywords: Epigenetic aging; Microbiome; Quality of Life; Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized crossover trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Delayed supplementation (Experimental): Participants will consume greens-based supplement for 30 days after living their normal lives (free-living) for 30 days.
  Interventions: Dietary Supplement: Greens-based Supplement
- Immediate supplementation (Experimental): Participant will consume greens-based supplement for 30 days after which they will crossover into a free-living/non-supplementation setting for 30 days.
  Interventions: Dietary Supplement: Greens-based Supplement

INTERVENTIONS:
Dietary Supplement: Greens-based Supplement — Participant will consume one serving of greens-based supplement per day in the morning, for 30 days.

SUMMARY:
The primary purpose of this study is to assess changes in epigenetic markers of aging and physiological parameters in overweight older adults consuming a mixed greens-based supplement over a 30-day period in a randomized crossover design.

DETAILED DESCRIPTION:
Investigators will recruit 20 overweight/obese but otherwise healthy participants aged 50-65. Participants will be randomized to consume the greens-based supplement each morning for the first 30 days or second 30 days of the study. Usual diet, physical activity, and sleep patterns will be encouraged and monitored during the duration of the study.

Phlebotomy will be conducted at baseline, 30-day crossover, and 60-day follow-up to assess DNA methylation in peripheral blood mononuclear cells. Visceral and total body fat, stool microbiome composition, and actigraphy will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of any ethnicity (women must be postmenopausal)
* Body Mass Index > 30 kg/m^2
* Low habitual dark green leafy vegetable consumption
* Willing to adhere to study protocol and measures
* Willing to communicate via smartphone technology
* Able to read, write and speak English

Exclusion Criteria:

* Overt cardiometabolic diseases such heart attack, stroke, diabetes, insulin resistance and non-alcoholic fatty liver disease, etc.
* Diagnosis of a transient ischemic attack in the 6 months prior to screening
* Diagnosis of cancer within 5 years prior to screening, except for cutaneous basal cell or squamous cell cancer resolved by excision
* Food allergies

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Changes in DNA Methylation in Peripheral Blood Mononuclear Cells | Change from day 0 (baseline) to day 30 post intervention supplementation.
  Change from Baseline in Epigenetic Aging Profiles (i.e. DNA Methylation), after 30 day intervention. Participants will provide blood samples at their baseline study visit, which occurs before the start of the intervention, and at their visit at the end of the 30th of intervention supplementation.

SECONDARY OUTCOMES:
Fasting serum triglycerides | Change from day 0 (baseline) to day 30 post intervention supplementation.
  Phlebotomy will be obtained while fasted 8+ hours and triglycerides will be measured as part of a comprehensive metabolic panel and reported in mg/dl. Lower concentrations are optimal.
Fasting serum low-density lipoproteins (LDL) | Change from day 0 (baseline) to day 30 post intervention supplementation.
  Phlebotomy will be obtained while fasted 8+ hours and low-density lipoproteins (LDL) will be measured as part of a comprehensive metabolic panel and reported in mg/dl. Lower concentrations are optimal.
Fasting serum blood glucose | Change from day 0 (baseline) to day 30 post intervention supplementation.
  Phlebotomy will be obtained while fasted 8+ hours and blood glucose will be measured as part of a comprehensive metabolic panel and reported in mg/dl. Lower concentrations are optimal.
Visceral fat percentage | Change from Day 0 (baseline), Day 30 (Crossover/Midpoint ), and Day 60 (end of study)
  Change in visceral fat as a percentage of total fat mass as measured by bioelectrical impedance (BIA). Lower values are optimal.
Total body fat percentage | Change from Day 0 (baseline), Day 30 (Crossover/Midpoint ), and Day 60 (end of study)
  Change in total body fat as a percentage of total fat mass as measured by bioelectrical impedance (BIA). Lower values are optimal.
Stool microbiome composition | Change from Day 0 (baseline), Day 30 (Crossover/Midpoint ), and Day 60 (end of study)
  16S changes in microbiome alpha diversity.
Breath Hydrogen (ppm) | Change from Day 0 (baseline), Day 30 (Crossover/Midpoint ), and Day 60 (end of study)
  Breath hydrogen will be measured via QuinTron BreathTracker SC Analyzer every 30 minutes to 1.5 hours on days 21 and 51. Lower levels are optimal.
Breath Methane (ppm) | Change from Day 0 (baseline), Day 30 (Crossover/Midpoint ), and Day 60 (end of study)
  Breath methane will be measured via QuinTron BreathTracker SC Analyzer every 30minutes to 1.5 hours on days 21 and 51. Lower levels are optimal.
Physical Quality of Life | Change from Baseline (day 0), Crossover/Midpoint (day 30), and End of study (day 60)
  The SF-12 PCS (Short Form-12, Physical Component Score) is a health-related quality of life measure that assesses general physical functioning and well-being. SF-12 PCS scores range from 0-100 with higher scores indicating better general physical health.
Sleep and Physical Activity- accelerometry | Change from Baseline (day 0), Crossover/Midpoint (day 30), and End of study (day 60)
  Average minutes of total daily sleep and physical activity measured via garmin watch.
Total caloric intake | Change from Baseline (day 0), Crossover/Midpoint (day 30), and End of study (day 60)
  Three 24-hour dietary recalls will be obtained and entered into the and analyzed in the Nutrition Data System for Research (NDSR).
Mental Quality of Life | Change from Baseline (day 0), Crossover/Midpoint (day 30), and End of study (day 60)
  The SF-12 MCS (Short Form-12, Mental Component Score) is a health-related quality of life measure that assesses general mental health status. SF-12 MCS scores range from 0-100 with higher scores indicating better general mental health.

CONTACTS AND LOCATIONS:
Overall Officials: MIchael D Roberts, PhD, Principal Investigator — Auburn University
Locations (1):
- Auburn University, Auburn, Alabama, United States